CLINICAL TRIAL: NCT03163186
Title: Transradial Versus Transfemoral Arterial Access for Transarterial Embolization Therapy of Hepatic Carcinoma: A Patient Outcomes, Satisfaction, and Cost Analysis
Brief Title: Transradial Versus Transfemoral Arterial Access in Liver Cancer Embolization: Randomized Trial to Assess Patient Outcomes and Satisfaction (BEST ACCESS Trial).
Acronym: ACCESS
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Ricardo Yamada, Assistant Professor, Division of Vascular and Interventional Radiology, Medical University of South Carolina
Other Study IDs: PRO33987
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Hepatic Carcinoma; Chemoembolizaton; Transarterial Embolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transarterial embolization — Transarterial hepatic embolization of liver cancer

SUMMARY:
To evaluate the safety, advantages, and appropriateness of performing transarterial hepatic emobolization of liver cancer via arterial access from the radial artery versus conventional transfemoral arterial access. The procedures that will be followed utilizing arterial access include transarterial chemoembolization (TACE), specifically performed for hepatocellular carcinoma, and transarterial embolization (TAE) which is performed for types of liver tumors such as carcinoid tumors or liver metastases.

DETAILED DESCRIPTION:
The use of transradial (TR) access for the purpose of diagnosis and intervention in the arterial system is a well-established concept, particularly in coronary angiography, with many distinct advantages over conventional transfemoral (TF) access. The first series of 100 coronary angiographic procedures performed via TR access, published by Campeau in 19891, demonstrated 88% technical success rate and a 6% asymptomatic radial artery occlusion rate. Further experience and data accumulated with the first TR angioplasty procedure in 1992 and the first TR coronary stent placement in 1993. TR access for coronary artery interventions in the United States has grown exponentially over the past few years with the proportion of transradial percutaneous coronary interventions (PCI) procedures increasing from 1.2% in the first quarter of 2007 to 16.1% in the third quarter of 20122. And yet, its usage is largely absent in the interventional radiology and vascular surgery communities.

Reasons for this include a lack of appropriate training and equipment, but the potential advantages of TR over TF access are abundant in both coronary and non-coronary applications. Firstly, the radial artery is more superficial than the femoral artery without surrounding neurovascular structures susceptible to injury. In addition, any sustained arterial damage is significantly less detrimental because of the hand's dual arterial vascular supply. In addition, the radial artery is readily compressible regardless of the patient's body habitus. This compressibility has been shown to decrease the incidence of post-procedural bleeding complications as well as cardiac mortality during PCI3,4,5. In addition to patient safety, there are numerous benefits to overall patient comfort and convenience. For one, after TR access, patients may sit up in bed and ambulate immediately with faster discharge to home. In one randomized trial, Cooper et al demonstrated a strong patient preference, improved quality-of-life metrics, and decreased hospital costs for TR over TF access during cardiac catherization6. These benefits have yet to be empirically demonstrated for non-coronary applications like transarterial hepatic embolization. Even so, these potential benefits are of even greater importance in the patient population undergoing chemoembolization/bland embolization given the chemo/bland embolization's association with nausea and emesis post intervention.

Ultimately, complications with TR approach have proven rare in both coronary and noncoronary applications. Most commonly, a local small hematoma may develop with mild pain, usually treated with NSAIDS if necessary. Despite meticulous hemostatic technique, radial artery thrombosis may occur. Nevertheless, this thrombosis almost always remains asymptomatic7, at least partially because a modified Allen's test is performed before all procedures using TR access. The Allen's test is a clincal examination technique that determines the presence of dual arterial supply to the hand and palmar arch patency in the event of radial artery occlusion. Additional possible complications of TR access include radial artery pseudoaneurysm, spasm, dissection, digit ischemia, as well as cerebral infarction, but all of the following have proven to be extremely low incidence particularly with the usage of intraprocedural heparinization and vasodilators, which are included in our procedure protocol.

Finally and increasing more importantly in the modern era of health care reform, TR access offers many benefits to hospital costs and patient satisfaction. Many studies have demonstrated decreased costs associated with TR versus traditional TF access5,8,9, primarily due to the nonutilization of arterial closure devices and decreased readmission for bleeding complications. International studies have long promoted TR access as a feasible, safe, and well tolerated method for performing hepatic transarterial chemoembolization10,11. In a recent series performed in the United States, technical success was obtained in all procedures. Furthermore, 100% of patients who underwent both TF and TR access preferred TR over TF access12. Our study seeks to further establish TR arterial access as a viable and typically preferable method for performing hepatic transarterial embolization as well as refine patient suitability criteria for TR access.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Selected for TACE treatment of Barcelona Clinic Liver Cancer Staging System stage B disease per current standard of care or TAE for the treatment of hepatic carcinoma
3. Radial diameter of ≥2.0mm as determined by clinical and ultrasound evaluation
4. Patient undergoes at least two of three courses of planned treatment with TACE/TAE per institutional protocol

Exclusion Criteria:

1. Need for additional procedures requiring transfemoral or transradial access approach during the same hospitalization
2. Patient is unable to give informed consent in accordance with guidelines established the Institutional Review Board.
3. Unsuitable for radial access due lack of dual arterial supply to the hand as determined by modified Allen test.
4. Female patients who are pregnant, breastfeeding, or premenopausal and not using an effective method of contraceptive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be patients referred to Division of Vascular Interventional Radiology (VIR) at MUSC found suitable for TACE per the Barcelona Clinic Liver Cancer Staging System with stage B disease (Eastern Cooperative Oncology Group (ECOG) performance status 0-2 and Child-Pugh A-B liver disease with or without portal vein thrombus). Our current institutional protocol to treat unresectable Hepatocellular Carcinoma(HCC) and hepatic metastatic includes three separate TACE/TAE procedures in average in order to obtain local tumor control.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2016-08-18 (Actual)

PRIMARY OUTCOMES:
To assess potential patient preference for the performance of hepatic embolization procedures via transradial versus transfemoral approach. | December, 2015 through August, 2016
  Record of patient response via administered questionnaire as well as stated patient choice in the selection of approach for the third planned procedure of a series. These findings will be correlated with additional objective data regarding complication rates.

SECONDARY OUTCOMES:
To evaluate complication rates and severity from different modes of access. | December, 2015 through August, 2016
  This data will be collected from imaging, clinical, and laboratory measures of complications collected at both the one day and follow-up clinic visits.
To assess ancillary procedural and patient satisfaction quality metrics between the two groups. | December, 2015 through August, 2016
  Procedural details include contrast amount, fluoroscopy time, operator exposure, and cost will also be collected and compared between the two treatment groups. Additional patient quality of life endpoints will be also be compared based on the results of items 1 through 7 on the post-procedure questionnaire.
To identify potential risk factors for complications in transradial approach. | December, 2015 through August, 2016
  This will be determined by evaluating association of complication data with pre-procedural laboratory and imaging evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States